CLINICAL TRIAL: NCT04747158
Title: COVID-19 Convalescent Plasma Therapy
Acronym: TPCC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Asunción (Other)
Collaborators: Consejo Nacional de Ciencias y Tecnología, Paraguay (Unknown); Ministerio de Salud Pública y Bienestar Social, Paraguay (Unknown); Centro de información y recursos para el desarrollo, Paraguay (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINV20-388
Record Dates: First submitted 2021-01-27; First posted 2021-02-10 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV-2 Infection; COVID-19 Infection
Keywords: SARS-CoV-2 infection; Convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent plasma (Experimental): COVID-19 convalescent plasma
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — COVID-19 convalescent plasma at admission, after confirmation of eligibility, 200 ml on day 1 and 2

SUMMARY:
This study is an open-label trial in which hospitalized patients with risk factors of severe coronavirus disease 2019 [COVID-19] will be receive treatment with convalescent plasma (≤ 15 days from symptoms start).

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Presence of risk factors of severe COVID 19 diagnosed by quantitative polymerase chain reaction by reverse transcription (RT-qPCR)
* Patients with no more than 15 days from the onset of symptoms
* Signed informed consent

Exclusion Criteria:

* Severely ill patients admitted directly to the ICU.
* Need for mechanical ventilation at the time of hospital admission, regardless of the time of clinical evolution.
* History of previous hypersensitivity to plasma transfusions.
* History of immunoglobulin A (IgA) deficiency
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Overall survival (30-day mortality) | 30 days
  To evaluate the effectiveness of convalescent plasma therapy COVID-19, to decrease mortality in hospitalized patients with COVID-19 and who present some risk factor for clinical deterioration.

SECONDARY OUTCOMES:
Median length of hospital stay | 30 days
  To describe the median length of hospital stay in days
Change in clinical status | 0, 3, 7 and 14 days
  To asses the changes of disease severity, according to the COVID-19 disease severity from the World Health Organization (WHO) Interim guidance.
Change in inflammatory marker: ferritin | 0, 7 and 14 days
  To measure changes in ferritin (μg/L) at 0, 7 and 14 days
Change in inflammatory marker: D dimer | 0, 7 and 14 days
  To measure changes in D dimer (mg/L) at 0, 7 and 14 days
Change in inflammatory marker: leukocytes | 0, 7 and 14 days
  To measure leukocytes (/mm3) changes at 0, 7 and 14 days
Serum Antibody Titers | 0, 3 and 7 days
  To measure immunoglobulin G (IgG) SARS-CoV 2 titles
Transfer to ICU | 30 days
  To asses the frequency of patients admitted to ICU
Transfusion related events | 4 hours
  To asses the frequency of adverse events to convalescent plasma

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Jimenez de Samudio, MD,MSc, Principal Investigator — Facultad de Ciencias Médicas - Universidad Nacional de Asunción
Locations (1):
- Facultad de Ciencias Médicas - Universidad Nacional de Asunción, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No
The investigators will publish the results to compare data with other studies with COVID-19 convalescent plasma patients

REFERENCES:
- [Background] Yoon HA, Bartash R, Gendlina I, Rivera J, Nakouzi A, Bortz RH 3rd, Wirchnianski AS, Paroder M, Fehn K, Serrano-Rahman L, Babb R, Sarwar UN, Haslwanter D, Laudermilch E, Florez C, Dieterle ME, Jangra RK, Fels JM, Tong K, Mariano MC, Vergnolle O, Georgiev GI, Herrera NG, Malonis RJ, Quiroz JA, Morano NC, Krause GJ, Sweeney JM, Cowman K, Allen S, Annam J, Applebaum A, Barboto D, Khokhar A, Lally BJ, Lee A, Lee M, Malaviya A, Sample R, Yang XA, Li Y, Ruiz R, Thota R, Barnhill J, Goldstein DY, Uehlinger J, Garforth SJ, Almo SC, Lai JR, Gil MR, Fox AS, Chandran K, Wang T, Daily JP, Pirofski LA. Treatment of Severe COVID-19 with Convalescent Plasma in the Bronx, NYC. medRxiv [Preprint]. 2020 Dec 4:2020.12.02.20242909. doi: 10.1101/2020.12.02.20242909. PMID 33300012
- [Background] Joyner MJ, Bruno KA, Klassen SA, Kunze KL, Johnson PW, Lesser ER, Wiggins CC, Senefeld JW, Klompas AM, Hodge DO, Shepherd JRA, Rea RF, Whelan ER, Clayburn AJ, Spiegel MR, Baker SE, Larson KF, Ripoll JG, Andersen KJ, Buras MR, Vogt MNP, Herasevich V, Dennis JJ, Regimbal RJ, Bauer PR, Blair JE, van Buskirk CM, Winters JL, Stubbs JR, van Helmond N, Butterfield BP, Sexton MA, Diaz Soto JC, Paneth NS, Verdun NC, Marks P, Casadevall A, Fairweather D, Carter RE, Wright RS. Safety Update: COVID-19 Convalescent Plasma in 20,000 Hospitalized Patients. Mayo Clin Proc. 2020 Sep;95(9):1888-1897. doi: 10.1016/j.mayocp.2020.06.028. Epub 2020 Jul 19. PMID 32861333
- [Background] Clinical Management of COVID-19 - Interim guidance 27 May 2020. WHO reference number: WHO/2019-nCoV/clinical/2020.5
- See also: Open data' page of projects funded by CONACYT, Paraguay — https://datos.conacyt.gov.py/proyectos/pdf/3449